CLINICAL TRIAL: NCT01702454
Title: Immunogenicity, Safety and Reactogenicity Study of GSK Biologicals' Quadrivalent Seasonal Influenza Candidate Vaccine GSK2321138A, Administered to Children Who Previously Participated in Study 115345
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Influenza Vaccine When Administered in Children Who Previously Participated in Study 115345
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116023; 2012-001230-34 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-07

CONDITIONS: Influenza
Keywords: GSK Biologicals quadrivalent influenza vaccine; Influenza; Children; Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Fluarix Quadrivalent Primed Group (Experimental): Subjects in this group were previously primed with 2 doses of Fluarix Quadrivalent vaccine in the primary study 115345 (NCT01439360) and received 1 dose of Fluarix Quadrivalent vaccine at Day 0 in the current study. The vaccine was administered intramuscularly in the deltoid region of arm.
  Interventions: Biological: Fluarix Quadrivalent
- Fluarix Quadrivalent Unprimed Group (Experimental): Subjects in this group were unprimed in the primary study 115345 (NCT01439360) and received 2 doses of Fluarix Quadrivalent vaccine at Days 0 and 28 in the current study. The vaccine was administered intramuscularly in the deltoid region of arm.
  Interventions: Biological: Fluarix Quadrivalent

INTERVENTIONS:
Biological: Fluarix Quadrivalent — 1 or 2 doses administered intramuscularly (IM) in deltoid region depending on the priming status

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of GSK Biologicals' investigational vaccine GSK2321138A in children who previously participated in study 115345 (FLU D-QIV-004 PRI) (NCT01439360).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/LAR(s) can and will comply with the requirements of the protocol.
* Children, male or female who received a 2-dose vaccination in the study 115345 (NCT01439360).
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Subjects in stable health as determined by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Since the start of study 115345 (NCT01439360), receipt of any seasonal influenza vaccine other than the study vaccines of study 115345 or planned administration of any influenza vaccine other than the study vaccine during the study.
* Administration of any vaccine not foreseen by the study protocol within 4 weeks preceding the first dose of study vaccine or planned use until Visit 2.
* Laboratory confirmed influenza infection outside of the 115345 (NCT01439360) study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to enrolment in the study or planned administration during the study period. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/ or any blood products within 3 months preceding the first dose of study vaccine or planned administration during the study period.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Any contraindication to intramuscular injection.
* Acute disease and/or fever at the time of enrollment:

  * Fever is defined as temperature ≥ 37.5°C by any route.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.

Ages: 17 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 470 (Actual)
Dates: Start 2012-10-06; Primary Completion 2013-05-06 (Actual); Study Completion 2013-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- Czechia (9):
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Lipník nad Bečvou
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Odolena Voda
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
- Poland (3):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Siemianowice Śląskie
- Spain (10):
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Blanes (Girona)
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Paiporta, Valencia
  - GSK Investigational Site, Quart de Poblet, Valencia
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- United Kingdom (9):
  - GSK Investigational Site, St Austell, Cornwall
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Gloucester
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Claeys C, Chandrasekaran V, Garcia-Sicilia J, Prymula R, Diez-Domingo J, Brzostek J, Mares-Bermudez J, Martinon-Torres F, Pollard AJ, Ruzkova R, Carmona Martinez A, Ulied A, Miranda Valdivieso M, Faust SN, Snape MD, Friel D, Ollinger T, Soni J, Schuind A, Li P, Innis BL, Jain VK. Anamnestic Immune Response and Safety of an Inactivated Quadrivalent Influenza Vaccine in Primed Versus Vaccine-Naive Children. Pediatr Infect Dis J. 2019 Feb;38(2):203-210. doi: 10.1097/INF.0000000000002217. PMID 30325891
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 116023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Started | 241 | 229
Completed | 238 | 221
Not Completed | 3 | 8
Not completed — Consent withdrawal | 0 | 1
Not completed — Migrated/moved from study area | 0 | 1
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group | Total
Number analyzed (Participants) | 241 | 229 | 470
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.2 (7.54) | 32.5 (7.39) | 32.8 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 96 | 210
  Male | 127 | 133 | 260

OUTCOME MEASURES:

1. Primary Outcome: Serum Hemagglutination Inhibition (HI) Antibody Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs). The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects who received study vaccine according to their treatment assignment, for whom assay results for antibodies against at least 1 study vaccine strain after vaccination and data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 224 | 209
Titer
  H1N1, Day 0 [N=221,202] | 43.1 [33.8 to 54.9] | 14.5 [11.5 to 18.2]
  H1N1, Day 7 [N=224,209] | 445.6 [376.9 to 526.7] | 45.8 [32.0 to 65.5]
  H3N2, Day 0 [N=221,202] | 12.3 [10.7 to 14.1] | 16.4 [13.2 to 20.4]
  H3N2, Day 7 [N=224,209] | 135.3 [113.6 to 161.2] | 47.5 [32.6 to 69.3]
  Victoria, Day 0 [N=221,202] | 28.5 [23.8 to 34.1] | 10.0 [8.4 to 11.9]
  Victoria, Day 7 [N=224,209] | 193.9 [168.7 to 222.8] | 47.1 [35.2 to 63.0]
  Yamagata, Day 0 [N=221,202] | 11.9 [10.6 to 13.3] | 6.5 [5.9 to 7.2]
  Yamagata, Day 7 [N=224,209] | 182.6 [159.0 to 209.6] | 26.1 [20.9 to 32.7]
Statistical Analysis 1: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; The adjusted GMT of HI antibodies for A/Christchurch strain at post-vaccination dose 1, the GMT ratio of Fluarix Quadrivalent Primed Group/Fluarix Quadrivalent Unprimed Group and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination log-10 titer and age as regressors; Test type: Non-Inferiority or Equivalence — Criterion: The lower limit (LL) of the two-sided 95% Confidence Interval (CI) for the GMT ratio is above 1; Adjusted GMT ratio = 8.97, 95% CI 2-sided [6.21 to 12.96] — The GMTs were used to calculate the Adjusted GMTs, which in turn were used to calculate the Adjusted GMT ratio with 95% confidence interval
Statistical Analysis 2: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; The adjusted GMT of HI antibodies for A/Victoria strain at post-vaccination dose 1, the GMT ratio of Fluarix Quadrivalent Primed Group/Fluarix Quadrivalent Unprimed Group and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination log-10 titer and age as regressors; Test type: Non-Inferiority or Equivalence — Criterion: The lower limit (LL) of the two-sided 95% Confidence Interval (CI) for the GMT ratio is above 1; Adjusted GMT ratio = 2.7, 95% CI 2-sided [1.81 to 4.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; The adjusted GMT of HI antibodies for B/Brisbane strain at post-vaccination dose 1, the GMT ratio of Fluarix Quadrivalent Primed Group/Fluarix Quadrivalent Unprimed Group and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination log-10 titer and age as regressors; Test type: Non-Inferiority or Equivalence — Criterion: The lower limit (LL) of the two-sided 95% Confidence Interval (CI) for the GMT ratio is above 1; Adjusted GMT ratio = 3.94, 95% CI 2-sided [2.89 to 5.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; The adjusted GMT of HI antibodies for B/Hub-Wuj strain at post-vaccination dose 1, the GMT ratio of Fluarix Quadrivalent Primed Group/Fluarix Quadrivalent Unprimed Group and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination log-10 titer and age as regressors; Test type: Non-Inferiority or Equivalence — Criterion: The lower limit (LL) of the two-sided 95% Confidence Interval (CI) for the GMT ratio is above 1; Adjusted GMT ratio = 6.71, 95% CI 2-sided [5.21 to 8.63] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Seropositive Subjects Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine
Description: Seropositivity was defined as number of subjects with antibody titers greater than or equal to (≥) 1:10. The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 224 | 209
Subjects
  H1N1, Day 0 [N=221,202] | 189 | 64
  H1N1, Day 7 [N=224,209] | 220 | 137
  H3N2, Day 0 [N=221,202] | 131 | 79
  H3N2, Day 7 [N=224,209] | 218 | 99
  Victoria, Day 0 [N=221,202] | 187 | 58
  Victoria, Day 7 [N=224,209] | 224 | 174
  Yamagata, Day 0 [N=221,202] | 134 | 36
  Yamagata, Day 7 [N=224,209] | 222 | 144

3. Primary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 7 post dose 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 221 | 202
Subjects
  H1N1 | 170 | 65
  H3N2 | 180 | 73
  Victoria | 169 | 78
  Yamagata | 208 | 77
Statistical Analysis 1: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; To assess the immune response in terms of SCR difference at Day 7 after one dose of Fluarix Quadrivalent vaccine (2012-2013 formulation) in vaccine-primed and vaccine-unprimed subjects, for all the strains; Test type: Non-Inferiority or Equivalence — SCR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in percentages = 44.74, 95% CI 2-sided [35.87 to 52.84]
Statistical Analysis 2: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — SCR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in percentages = 45.31, 95% CI 2-sided [36.58 to 53.3]
Statistical Analysis 3: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — SCR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in percentages = 37.86, 95% CI [28.83 to 46.26]
Statistical Analysis 4: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; To assess the immune response in terms of SCR difference at Day 7 after one dose of Fluarix Quadrivalent vaccine (2012-2013 formulation) in vaccine-primed and vaccine-unprimed subjects, for all the strains. B/Hu-Wuj = B/Hubei-Wujiagang/158/2009 (Yamagata); Test type: Non-Inferiority or Equivalence — SCR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in percentages = 56, 95% CI [48.32 to 63.04]

4. Primary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titer Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: MGI was defined as the fold increase in serum HI GMT post-vaccination compared to Day 0. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 7 post dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 221 | 202
Fold increase
  H1N1 | 10.3 [8.5 to 12.4] | 3.2 [2.6 to 3.9]
  H3N2 | 10.9 [9.4 to 12.6] | 2.9 [2.4 to 3.6]
  Victoria | 6.7 [5.9 to 7.6] | 4.6 [3.8 to 5.5]
  Yamagata | 15.2 [13.3 to 17.3] | 4.0 [3.3 to 4.9]

5. Primary Outcome: Number of Subjects Seroprotected for Anti-HA Antibodies Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: Seroprotection rate (SPR) was defined as the number of vaccinees with serum haemagglutination inhibition (HI) titer ≥ 1:40 that usually is accepted as indicating protection in adults. The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 224 | 209
Subjects
  H1N1, Day 0 [N=221,202] | 89 | 61
  H1N1, Day 7 [N=224,209] | 217 | 72
  H3N2, Day 0 [N=221,202] | 37 | 74
  H3N2, Day 7 [N=224,209] | 193 | 81
  Victoria, Day 0 [N=221,202] | 72 | 39
  Victoria, Day 7 [N=224,209] | 217 | 84
  Yamagata, Day 0 [N=221,202] | 27 | 12
  Yamagata, Day 7 [N=224,209] | 216 | 83
Statistical Analysis 1: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; To assess the immune response in terms of SPR difference at Day 7 after one dose of Fluarix Quadrivalent vaccine (2012-2013 formulation) in vaccine-primed and vaccine-unprimed subjects, for all the strains; Test type: Non-Inferiority or Equivalence — SPR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in SPR = 62.43, 95% CI 2-sided [55.27 to 68.89]
Statistical Analysis 2: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — SPR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in SPR = 47.4, 95% CI 2-sided [39.08 to 55.06]
Statistical Analysis 3: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — SPR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in SPR = 56.68, 95% CI 2-sided [49.44 to 63.43]
Statistical Analysis 4: Comparison: Fluarix Quadrivalent Primed Group vs Fluarix Quadrivalent Unprimed Group; To assess the immune response in terms of SPR difference at Day 7 after one dose of Fluarix Quadrivalent vaccine (2012-2013 formulation) in vaccine-primed and vaccine-unprimed subjects, for all the strains. B/Hu-Wuj = B/Hubei-Wujiagang/158/2009 (Yamagata); Test type: Non-Inferiority or Equivalence — SPR difference was calculated using standardized asymptotic 95% CI for the group difference in proportion; Difference in SPR = 56.72, 95% CI 2-sided [49.41 to 63.49]

6. Primary Outcome: Serum Hemagglutination Inhibition (HI) Antibody Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: as for outcome 1
Time Frame: At Day 0 and Day 7
Population: Analyses was performed on According-to-Protocol cohort for immunogenicity (ATP-I) excluding subjects who had an RT-PCR confirmed influenza infection in study 115345 consisted of all evaluable subjects from the ATP-I, excluding subjects who had an RT-PCR confirmed influenza infection in study 115345.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Fluarix Quadrivalent Primed Group: Subjects in this group were previously primed with 2 doses of Fluarix Quadrivalent vaccine in the primary study 115345 (NC T01439360) and received 1 dose of Fluarix Quadrivalent vaccine at Day 0 in the current study. The vaccine was administered intramuscularly in the deltoid region of arm.
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 213 | 179
Titers
  H1N1, Day 0 [N=210,173] | 44.0 [34.2 to 56.7] | 14.3 [11.2 to 18.3]
  H1N1, Day 7 [N=213,179] | 442.3 [372.0 to 525.9] | 42.7 [29.0 to 63.0]
  H3N2, Day 0 [N=210,173] | 11.0 [9.8 to 12.5] | 11.9 [9.6 to 14.7]
  H3N2, Day 7 [N=213,179] | 125.9 [105.4 to 150.4] | 28.7 [19.7 to 41.9]
  Victoria, Day 0 [N=210,173] | 27.8 [23.2 to 33.2] | 10.3 [8.5 to 12.5]
  Victoria, Day 7 [N=213,179] | 193.3 [167.6 to 222.8] | 46.1 [33.5 to 63.4]
  Yamagata, Day 0 [N=210,173] | 11.9 [10.6 to 13.4] | 6.5 [5.8 to 7.2]
  Yamagata, Day 7 [N=213,179] | 184.1 [159.8 to 212.1] | 25.2 [19.8 to 32.0]

7. Primary Outcome: Number of Subjects Seropositive for HI Antibody Titers Against Each of the Four Vaccine Strains After Dose 1 of Fluarix Quadrivalent Vaccine
Description: as for outcome 2
Time Frame: At Day 0 and Day 7
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 213 | 179
Subjects
  H1N1, Day 0 [N=210,173] | 178 | 54
  H1N1, Day 7 [N=213,179] | 209 | 113
  H3N2, Day 0 [N=210,173] | 120 | 52
  H3N2, Day 7 [N=213,179] | 207 | 72
  Victoria, Day 0[ N=210,173] | 177 | 50
  Victoria, Day 7[ N=213,179] | 213 | 145
  Yamagata, Day 0[ N=210,173] | 127 | 31
  Yamagata, Day 7 [N=213,179] | 211 | 120

8. Primary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a four-fold increase in post-vaccination titer. The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria)and B/Hubei-Wujiagang/158/2009 (Yamagata )antigens.
Time Frame: At Day 7 post dose 1
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 210 | 173
Subjects
  H1N1, Day 7 [N=210,173] | 160 | 54
  H3N2, Day 7 [N=210,173] | 173 | 49
  Victoria, Day 7 [N=210,173] | 162 | 66
  Yamagata, Day 7 [N=210,173] | 197 | 65

9. Primary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: Mean geometric increase was defined as the geometric mean of the within subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011(H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 7 post dose 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 210 | 173
Fold Increase
  H1N1, Day 7 [N=210,173] | 10.0 [8.1 to 12.2] | 3.1 [2.5 to 3.9]
  H3N2, Day 7 [N=210,173] | 11.2 [9.7 to 13.1] | 2.4 [2.0 to 3.0]
  Victoria, Day 7 [N=210,173] | 6.9 [6.0 to 7.8] | 4.5 [3.7 to 5.4]
  Yamagata, Day 7 [N=210,173] | 15.2 [13.3 to 17.4] | 4.0 [3.2 to 4.9]

10. Primary Outcome: Number of Subjects Seroprotected for HI Antibodies Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: Seroprotection rate was defined as the number of vaccinees with a serum HI titer greater than or equal to(≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011(H3N2), B/Brisbane/60/2008 (Victoria)and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 213 | 179
Subjects
  H1N1,Day 0 [N=210,173] | 87 | 51
  H1N1, Day 7 [N=213,179] | 206 | 59
  H3N2, Day 0 [N=210,173] | 29 | 48
  H3N2, Day 7 [N=213,179] | 182 | 54
  Victoria, Day 0 [N=210,173] | 68 | 35
  Victoria, Day 7 [N=213,179] | 206 | 70
  Yamagata, Day 0 [N=210,173] | 27 | 10
  Yamagata, Day 7 [N=213,179] | 205 | 70

11. Secondary Outcome: Number of Subjects With HI Antibody Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: The cut-off values assessed were less than (<) 1:10, 1:10 to < 1:40 and ≥ 1:40. The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 224 | 209
Subjects
  H1N1 (<1:10), Day 0 [N=221,202] | 32 | 138
  H1N1 (<1:10), Day 7 [N=224,209] | 4 | 72
  H3N2 (<1:10), Day 0 [N=221,202] | 90 | 123
  H3N2 (<1:10), Day 7 [N=224,209] | 6 | 110
  Victoria (<1:10), Day 0 [N=221,202] | 34 | 144
  Victoria (<1:10), Day 7 [N=224,209] | 0 | 35
  Yamagata (<1:10), Day 0 [N=221,202] | 87 | 166
  Yamagata (<1:10), Day 7 [N=224,209] | 2 | 65
  H1N1 (1:10 to <1:40), Day 0 [N=221,202] | 100 | 3
  H1N1 (1:10 to <1:40), Day 7 [N=224,209] | 3 | 65
  H3N2 (1:10 to <1:40), Day 0 [N=221,202] | 94 | 5
  H3N2 (1:10 to <1:40), Day 7 [N=224,209] | 25 | 18
  Victoria (1:10 to <1:40), Day 0 [N=221,202] | 115 | 19
  Victoria (1:10 to <1:40), Day 7 [N=224,209] | 7 | 90
  Yamagata (1:10 to <1:40), Day 0 [N=221,202] | 107 | 24
  Yamagata (1:10 to <1:40), Day 7 [N=224,209] | 6 | 61
  H1N1 (≥1: 40), Day 0 [N=221,202] | 89 | 61
  H1N1 (≥1: 40), Day 7 [N=224,209] | 217 | 72
  H3N2 (≥1: 40), Day 0 [N=221,202] | 37 | 74
  H3N2 (≥1: 40), Day 7 [N=224,209] | 193 | 81
  Victoria (≥1: 40), Day 0 [N=221,202] | 72 | 39
  Victoria (≥1: 40), Day 7 [N=224,209] | 217 | 84
  Yamagata (≥1: 40), Day 0 [N=221,202] | 27 | 12
  Yamagata (≥1: 40), Day 7 [N=224,209] | 216 | 83

12. Secondary Outcome: Serum Neutralising Antibody Titers Against Each of the Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine
Description: as for outcome 1
Time Frame: At Day 0 and Day 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 107 | 109
Titer
  H1N1, Day 0 [N=97,90] | 138.2 [97.4 to 196.2] | 48.3 [33.9 to 68.7]
  H1N1, Day 7 [N=107, 96] | 1500.9 [1172.7 to 1920.9] | 139.4 [78.8 to 246.8]
  H3N2, Day 0 [N=99,96] | 66.5 [55.9 to 79.2] | 82.8 [60.6 to 113.1]
  H3N2, Day 7 [N=104,100] | 422.9 [342.3 to 522.4] | 325.1 [187.1 to 564.7]
  Victoria, Day 0 [N=107,109] | 38.6 [29.7 to 50.3] | 22.2 [18.6 to 26.5]
  Victoria, Day 7 [N=107, 108] | 193.7 [154.7 to 242.6] | 47.0 [30.3 to 72.9]
  Yamagata, Day 0 [N=107,107] | 36.9 [34.2 to 39.8] | 30.8 [29.0 to 32.6]
  Yamagata, Day 7 [N=107,107] | 182.7 [157.7 to 211.8] | 51.7 [42.2 to 63.4]

13. Secondary Outcome: Serum Anti-neuraminidase Antibody Titers Against Each of the Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine
Description: Antibody titers were expressed as GMTs. The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 107 | 109
Titer
  H1N1, Day 0 [N=106,106] | 34.6 [25.3 to 47.3] | 24.1 [18.6 to 31.1]
  H1N1, Day 7 [N=106, 109] | 293.9 [247.2 to 349.3] | 41.3 [28.9 to 59.0]
  H3N2, Day 0 [N=107,106] | 38.4 [33.7 to 43.7] | 58.8 [47.2 to 73.4]
  H3N2, Day 7 [N=107, 109] | 189.4 [155.9 to 230.2] | 114.2 [84.1 to 155.2]
  Victoria, Day 0 [N=106,106] | 17.4 [14.2 to 21.3] | 14.3 [12.4 to 16.5]
  Victoria, Day 7 [N=106,109] | 90.6 [74.1 to 110.8] | 27.6 [19.4 to 39.1]
  Yamagata, Day 0 [N=106, 106] | 25.3 [21.6 to 29.6] | 15.4 [13.2 to 18.0]
  Yamagata, Day 7 [N=106,109] | 222.0 [185.7 to 265.4] | 40.6 [29.5 to 55.7]

14. Secondary Outcome: Vaccine Response Rate (VRR) for Neutralising Antibody Titers Against Each of the Four Vaccine Strains.
Description: VRR was defined as the number of vaccinees who had either a pre-vaccination titer <cut-off and a post-vaccination titer ≥ 4-fold of half of the cut-off or a pre-vaccination titer ≥cut-off and at least a 4-fold increase in post-vaccination titers. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 7 post dose 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 107 | 108
Subjects
  H1N1 [N=97,89] | 74 | 36
  H3N2 [N=97,94] | 72 | 48
  Victoria [N=107,108] | 78 | 24
  Yamagata [N=107,105] | 45 | 15

15. Secondary Outcome: MGI for Neutralising Antibodies Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: as for outcome 4
Time Frame: At Day 7 post dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 107 | 108
Fold increase
  H1N1 [N=97, 89] | 10.6 [8.2 to 13.7] | 3.1 [2.3 to 4.2]
  H3N2 [N=97, 94] | 6.4 [5.4 to 7.6] | 4.5 [3.2 to 6.2]
  Victoria [N=107,108] | 5.0 [4.3 to 5.8] | 2.1 [1.6 to 2.8]
  Yamagata [N=107,105] | 5.0 [4.3 to 5.7] | 1.7 [1.4 to 2.0]

16. Secondary Outcome: Vaccine Response Rate(VRR) for Anti-neuraminidase Antibody Titers Against Each of the Four Vaccine Strains.
Description: as for outcome 14
Time Frame: At Day 7 post dose 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 107 | 106
Subjects
  H1N1 [N=105,106] | 75 | 31
  H3N2 [N=107,106] | 75 | 31
  Victoria [N=105,106] | 79 | 24
  Yamagata [N=105,106] | 90 | 29

17. Secondary Outcome: MGI for Anti-neuraminidase Antibodies Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: as for outcome 4
Time Frame: At Day 7 post dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 107 | 106
Fold increase
  H1N1 [N=105,106] | 8.3 [6.5 to 10.7] | 1.8 [1.5 to 2.1]
  H3N2 [N=105,106] | 5.2 [4.4 to 6.0] | 1.9 [1.5 to 2.4]
  Victoria [N=105,106] | 8.8 [7.5 to 10.2] | 2.7 [2.1 to 3.4]
  Yamagata [N=107,106] | 4.9 [4.2 to 5.8] | 2.0 [1.7 to 2.3]

18. Secondary Outcome: Number of Subjects With HI Antibody Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: The cut-off values assessed were less than (<) 1:10, 1:10 to < 1:40,≥ 1:40, ≥1:60 and ≥1:80 . The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 213 | 179
Subjects
  H1N1, Day 0, <1:10 [N=210,173] | 32 | 119
  H1N1, Day 7, <1:10 [N=213,179] | 4 | 66
  H1N1, Day 0, 1:10 to <1:40 [N=210,173] | 178 | 54
  H1N1, Day 7, 1:10 to <1:40 [N=213,179] | 209 | 113
  H1N1, Day 0, ≥1:40 [N=210,173] | 87 | 51
  H1N1, Day 7, ≥1:40 [N=213,179] | 206 | 59
  H1N1, Day 0, ≥1:60 [N=210,173] | 73 | 47
  H1N1, Day 7, ≥1:60 [N=213,179] | 204 | 57
  H1N1, Day 0, ≥1:80 [N=210,173] | 73 | 47
  H1N1, Day 7, ≥1:80 [N=213,179] | 204 | 57
  H3N2, Day 0, <1:10 [N=210,173] | 90 | 121
  H3N2, Day 7, <1:10 [N=213,179] | 6 | 107
  H3N2, Day 0,1:10 to 1:40 [N=210,173] | 120 | 52
  H3N2, Day 7,1:10 to 1:40 [N=213,179] | 207 | 72
  H3N2, Day 0, ≥1:40 [N=210,173] | 29 | 48
  H3N2, Day 7, ≥1:40 [N=213,179] | 182 | 54
  H3N2, Day 0, ≥1:60 [N=210,173] | 12 | 36
  H3N2, Day 7, ≥1:60 [N=213,179] | 147 | 52
  H3N2, Day 0, ≥1:80 [N=210,173] | 12 | 36
  H3N2, Day 7, ≥1:80 [N=213,179] | 147 | 52
  Victoria, Day 0, <1:10 [N=210,173] | 33 | 123
  Victoria, Day 7, <1:10 [N=213,179] | 0 | 34
  Victoria, Day 0,1:10 to 1:40 [N=210,173] | 177 | 50
  Victoria, Day 7,1:10 to 1:40 [N=213,179] | 213 | 145
  Victoria, Day 0, ≥1:40 [N=210,173] | 68 | 35
  Victoria, Day 7, ≥1:40 [N=213,179] | 206 | 70
  Victoria, Day 0, ≥1:60 [N=210,173] | 40 | 27
  Victoria, Day 7, ≥1:60 [N=213,179] | 182 | 51
  Victoria, Day 0, ≥1:80 [N=210,173] | 40 | 27
  Victoria, Day 7, ≥1:80 [N=213,179] | 182 | 51
  Yamagata, Day 0, <1:10 [N=210,173] | 83 | 142
  Yamagata, Day 7, <1:10 [N=213,179] | 2 | 59
  Yamagata, Day 0,1:10 to 1:40 [N=210,173] | 127 | 31
  Yamagata, Day 7,1:10 to 1:40 [N=213,179] | 211 | 120
  Yamagata, Day 0, ≥1:40 [N=210,173] | 27 | 10
  Yamagata, Day 7, ≥1:40 [N=213,179] | 205 | 70
  Yamagata, Day 0, ≥1:60 [N=210,173] | 7 | 4
  Yamagata, Day 7, ≥1:60 [N=213,179] | 177 | 44
  Yamagata, Day 0, ≥1:80 [N=210,173] | 7 | 4
  Yamagata, Day 7, ≥1:80 [N=213,179] | 177 | 44

19. Secondary Outcome: Serum Micro Neutralizing(MN) Antibody Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: MN antibody titers were expressed as geometric mean titers(GMTs). The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 100 | 89
Titer
  H1N1,Day 0[N=90,72] | 141.4 [97.6 to 205.0] | 47.3 [32.1 to 69.6]
  H1N1,Day 7[N=100,76] | 1461.3 [1132.8 to 1885.1] | 138.4 [71.9 to 266.4]
  H3N2,Day 0[N=92,76] | 60.0 [51.2 to 70.4] | 59.6 [42.5 to 83.7]
  H3N2,Day 7[N=97,80] | 374.6 [305.4 to 459.4] | 177.7 [97.4 to 324.2]
  Victoria,Day 0[N=100,89] | 37.1 [28.6 to 48.2] | 23.5 [19.1 to 28.9]
  Victoria,Day 7[N=100,88] | 189.9 [151.2 to 238.5] | 52.0 [31.3 to 86.3]
  Yamagata,day 0[N=100,87] | 37.1 [34.2 to 40.2] | 30.9 [28.9 to 32.9]
  Yamagata, Day 7[N=100,88] | 177.5 [154.2 to 204.5] | 49.8 [40.5 to 61.1]

20. Secondary Outcome: Serum Anti-neuraminidase Antibody Titers Against Each of the Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine
Description: NI (Neuraminidase inhibitor) antibody titers were expressed as geometric mean titers(GMTs).The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 0 and Day 7
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 100 | 89
Titer
  H1N1, Day 0[N=99,86] | 34.8 [25.1 to 48.1] | 23.5 [17.8 to 31.1]
  H1N1, Day 7[N=99,89] | 287.1 [239.8 to 343.6] | 38.3 [25.7 to 57.1]
  H3N2, Day 0[N=100,86] | 35.0 [31.3 to 39.1] | 45.9 [36.7 to 57.4]
  H3N2, Day 7[N=100,89] | 175.8 [143.9 to 214.7] | 84.5 [60.7 to 117.6]
  Victoria, Day 0[N=99,86] | 16.8 [13.7 to 20.7] | 15.0 [12.7 to 17.6]
  Victoria, Day 7[N=99,89] | 89.2 [72.5 to 109.7] | 29.1 [19.6 to 43.2]
  Yamagata, Day 0[N=99,86] | 25.1 [21.3 to 29.5] | 15.4 [12.9 to 18.3]
  Yamagata, Day 7[N=100,89] | 216.5 [180.5 to 259.6] | 39.7 [27.9 to 56.6]

21. Secondary Outcome: Vaccine Response Rate(VRR) for Serum Neutralising Antibody Titers Against Each of the Four Vaccine Strains
Description: as for outcome 14
Time Frame: At Day 7 post dose 1
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 100 | 88
Subjects
  H1N1, Day 7[N=90,71] | 67 | 28
  H3N2, Day 7[N=90,74] | 66 | 31
  Victoria, Day 7[N=100,88] | 74 | 21
  Yamagata, Day 7[N=100,86] | 42 | 11

22. Secondary Outcome: MGI for Neutralising Antibodies Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine.
Description: MGI was defined as the fold increase in GMTs post-vaccination compared to Day 0. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 7 post dose 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 100 | 88
Fold Increase
  H1N1, Day 7[N=90,71] | 10.0 [7.7 to 13.1] | 3.1 [2.2 to 4.3]
  H3N2, Day 7[N=90,74] | 6.2 [5.2 to 7.5] | 3.4 [2.4 to 4.9]
  Victoria, Day 7[N=100,88] | 5.1 [4.4 to 5.9] | 2.2 [1.6 to 3.0]
  Yamagata, Day 7[N=100,86] | 4.8 [4.2 to 5.4] | 1.6 [1.3 to 1.9]

23. Secondary Outcome: Vaccine Response Rate(VRR) for Anti-neuraminidase Antibodies Against Each of the Four Vaccine Strains.
Description: VRR was defined as the percentage of vaccinees who had either a pre-vaccination titer <cut-off and a post-vaccination titer ≥ 4-fold of half of the cut-off or a pre-vaccination titer ≥cut-off and at least a 4-fold increase in post-vaccination titers. The vaccine strains included A/Christchurch/16/2010 ( H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.
Time Frame: At Day 7 post dose 1
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 100 | 86
Subjects
  H1N1, Day 7[N=98,86] | 70 | 23
  H3N2, Day 7[N=100,86] | 70 | 22
  Victoria, Day 7[N=98,86] | 74 | 20
  Yamagata, Day 7[N=99,86] | 85 | 23

24. Secondary Outcome: MGI for Anti-neuraminidase Antibodies Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine
Description: as for outcome 22
Time Frame: At Day 7 post dose 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 100 | 86
Fold increase
  H1N1, Day 7[N=98,86] | 8.1 [6.2 to 10.5] | 1.7 [1.4 to 2.1]
  H3N2, Day 7[N=100,86] | 5.0 [4.2 to 6.0] | 1.8 [1.6 to 2.2]
  Victoria, Day 7[N=98,86] | 5.2 [4.5 to 6.1] | 1.9 [1.5 to 2.5]
  Yamagata, Day 7[N=99,86] | 8.7 [7.4 to 10.2] | 2.6 [2.0 to 3.5]

25. Secondary Outcome: Serum Neutralising Antibody Titers Against Each of the Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine by Age Strata.
Description: Antibody titers were expressed as geometric mean titers. The vaccine strains included A/Christchurch/16/2010 (H1N1),A/Victoria/361/2011 (H3N2), A/Victoria/361/2011 and B/Hubei-Wujiagang/158/2009)(Yamagata) antigens. The humoral response in terms of neutralising antibodies for all vaccine strains were calculated by age stratum which included 17-29 months and 30-48 months age groups for both the Fluarix primed and unprimed groups.
Time Frame: At Day 0 and Day 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 54 | 55
Titers
  H1N1, Day 0,17-29M[N=47,44] | 76.8 [48.8 to 120.9] | 29.0 [18.7 to 44.9]
  H1N1, Day 7,17-29M [N=53,48] | 1112.0 [746.0 to 1657.8] | 53.0 [26.9 to 104.2]
  H1N1, Day 0,30-48M[N=50,46] | 240.0 [146.2 to 394.1] | 78.8 [46.6 to 133.1]
  H1N1, Day 7,30-48M[N=54,48] | 2014.5 [1517.5 to 2674.4] | 366.9 [155.6 to 865.4]
  H3N2,Day 0,17-29M[N=49,47] | 58.1 [46.3 to 72.9] | 74.5 [45.8 to 121.5]
  H3N2,Day 7,17-29M[N=51,50] | 370.5 [272.7 to 503.2] | 217.5 [97.0 to 488.0]
  H3N2,Day 0,30-48M[N=50,49] | 76.0 [58.2 to 99.1] | 91.5 [60.8 to 137.7]
  H3N2,Day 7,30-48M[N=53,50] | 480.3 [356.7 to 646.8] | 485.8 [226.2 to 1043.7]
  Victoria,Day 0,17-29M[N=53,54] | 29.2 [21.7 to 39.2] | 19.8 [15.9 to 24.8]
  Victoria,Day 7,17-29M[N=53,53] | 156.3 [119.7 to 204.2] | 35.5 [20.0 to 62.9]
  Victoria,Day 0,30-48M[N=54,55] | 50.9 [33.1 to 78.2] | 24.7 [18.8 to 32.6]
  Victoria,Day 7,30-48M[N=54,55] | 239.1 [166.7 to 343.0] | 61.8 [31.6 to 120.8]
  Yamagata, Day 0,17-29M[N=53,53] | 35.6 [32.3 to 39.2] | 29.6 [28.0 to 31.4]
  Yamagata, Day 7,17-29M[N=53,52] | 156.9 [129.4 to 190.3] | 45.6 [33.7 to 61.7]
  Yamagata, Day 0,30-48M[N=54,54] | 38.3 [34.0 to 43.1] | 32.0 [28.9 to 35.4]
  Yamagata, Day 7,30-48M[N=54,55] | 212.2 [170.1 to 264.7] | 58.3 [44.1 to 77.0]

26. Secondary Outcome: Serum Anti-neuraminidase Antibody Titers Against Each of the Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine by Age Strata
Description: Antibody titers were expressed as geometric mean titers. The vaccine strains included A/Christchurch/16/2010(H1N1), A/Victoria/361/2011(H3N2),B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009(Yamagata) antigens. The humoral response in terms of anti-neuraminidase antibodies for all vaccine strains were calculated by age stratum which included 17-29 months and 30-48 months age groups for both the Fluarix primed and unprimed groups.
Time Frame: At Day 0 and Day 7
Population: Analyses were performed on the ATP cohort for immunogenicity which included all evaluable subjects who received the study vaccine according to their treatment assignment, for whom the assay results for antibodies against at least one study vaccine strain after vaccination and for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 54 | 55
Titers
  H1N1, Day 0,17-29M[N=53,52] | 21.6 [15.0 to 31.3] | 15.8 [11.9 to 21.1]
  H1N1, Day 7,17-29M[N=53,54] | 246.3 [189.1 to 320.8] | 22.9 [14.9 to 35.1]
  H1N1, Day 0,30-48M[N=53,54] | 55.5 [34.2 to 89.9] | 36.1 [24.2 to 53.9]
  H1N1, Day 7,30-48M[N=53,55] | 350.7 [281.1 to 437.4] | 73.7 [42.9 to 126.7]
  H3N2, Day 0,17-29M[N=53,52] | 34.7 [29.2 to 41.2] | 49.8 [35.9 to 69.3]
  H3N2, Day 7,17-29M[N=53,54] | 158.0 [117.8 to 211.8] | 85.3 [55.4 to 131.4]
  H3N2, Day 0,30-48M[N=54,54] | 42.4 [34.9 to 51.6] | 69.0 [51.1 to 93.2]
  H3N2, Day 7,30-48M[N=54,55] | 226.4 [174.9 to 292.9] | 152.2 [98.5 to 235.1]
  Victoria, Day 0,17-29M[N=53,52] | 13.2 [11.0 to 16.0] | 13.1 [10.9 to 15.7]
  Victoria, Day 7,17-29M[N=53,54] | 68.8 [53.3 to 88.9] | 21.1 [13.4 to 33.2]
  Victoria, Day 0,30-48M[N=53,54] | 22.8 [16.0 to 32.4] | 15.7 [12.6 to 19.4]
  Victoria, Day 7,30-48M[N=53,55] | 119.2 [88.2 to 161.1] | 35.9 [21.0 to 61.4]
  Yamagata, Day 0,17-29M[N=53,52] | 20.5 [16.9 to 24.9] | 13.2 [11.1 to 15.8]
  Yamagata, Day 7,17-29M[N=53,54] | 181.4 [143.3 to 229.5] | 29.3 [19.5 to 44.0]
  Yamagata, Day 0,30-48M[N=53,54] | 31.1 [24.4 to 39.7] | 17.9 [13.8 to 23.1]
  Yamagata, Day 7,30-48M[N=53,55] | 271.8 [208.6 to 354.3] | 55.8 [34.4 to 90.5]

27. Secondary Outcome: Vaccine Response Rate(VRR) for Serum Neutralising Antibody Titers Against Each of the Four Vaccine Strains by Age Strata
Description: VRR was defined as the percentage of vaccinees who had either a pre-vaccination titer <cut-off and a post-vaccination titer ≥ 4-fold of half of the cut-off or a pre-vaccination titer ≥cut-off and at least a 4-fold increase in post-vaccination titers. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011(H3N2), B/Brisbane/60/2008(Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens. The humoral response in terms of neutralising antibodies for all vaccine strains were calculated by age stratum which included 17-29 months and 30-48 months age groups for both the Fluarix primed and unprimed groups.
Time Frame: At Day 7 post dose 1
Population: Analyses were perfomed on the ATP cohort for immunogenicity which included all evaluable subjects who received the study vaccine according to their treatment assignment, for whom the assay results for antibodies against at least one study vaccine strain after vaccination and for whom data concerning immunogenicity outcome measures were available
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 54 | 55
Subjects
  H1N1, Day 7, 17-29M[47,44] | 39 | 12
  H1N1, Day 7, 30-48M[50,45] | 35 | 24
  H3N2, Day 7,17-29M[N=48,46] | 36 | 19
  H3N2, Day 7,30-48M[N=49,48] | 36 | 29
  Victoria, Day 7,17-29M[N=53,53] | 41 | 9
  Victoria, Day 7,30-48M[N=54,55] | 37 | 15
  Yamagata, Day 7,17-29M[N=53,51] | 17 | 6
  Yamagata, Day 7,30-48M[N=54,54] | 28 | 9

28. Secondary Outcome: MGI for Neutralising Antibodies Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine by Age Strata
Description: MGI was defined as the fold increase in GMTs post-vaccination compared to Day 0.The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens.The humoral response in terms of neutralising antibodies for all vaccine strains were calculated by age stratum which included 17-29 months and 30-48 months age groups for both the Fluarix primed and unprimed groups.
Time Frame: At Day 7 post dose 1
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 54 | 55
Fold Increase
  H1N1, Day 7, 17-29M[N=47,44] | 13.1 [9.2 to 18.8] | 2.0 [1.4 to 3.0]
  H1N1, Day 7, 30-48M[N=50,45] | 8.7 [6.0 to 12.5] | 4.7 [3.0 to 7.3]
  H3N2, Day 7,17-29M[N=48,46] | 6.1 [4.8 to 7.7] | 3.4 [2.1 to 5.4]
  H3N2, Day 7,30-48M[N=49,48] | 6.7 [5.1 to 8.8] | 5.9 [3.8 to 9.2]
  Victoria, Day 7,17-29M[N=53,53] | 5.4 [4.4 to 6.5] | 1.8 [1.2 to 2.6]
  Victoria, Day 7,30-48M[N=54,55] | 4.7 [3.8 to 5.8] | 2.5 [1.6 to 3.8]
  Yamagata, Day 7,17-29M[N=53,51] | 4.4 [3.8 to 5.2] | 1.5 [1.2 to 2.0]
  Yamagata, Day 7,30-48M[N=54,54] | 5.5 [4.5 to 6.9] | 1.8 [1.4 to 2.4]

29. Secondary Outcome: Vaccine Response Rate(VRR) for Anti-neuraminidase Antibody Titers Against Each of the Four Vaccine Strains by Age Strata.
Description: VRR was defined as the percentage of vaccinees who had either a pre-vaccination titer <cut-off and a post-vaccination titer ≥ 4-fold of half of the cut-off or a pre-vaccination titer ≥cut-off and at least a 4-fold increase in post-vaccination titers. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria /361/2011(H3N2), B/Brisbane /60/2008(Victoria ) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens. The humoral response in terms of anti-neuraminidase antibodies for all vaccine strains were calculated by age stratum which included 17-29 months and 30-48 months age groups for both the Fluarix primed and unprimed groups.
Time Frame: At Day 7 post dose 1
Population: as for outcome 26
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 54 | 54
Subjects
  H1N1, Day 7,17-29M[N=53,52] | 43 | 11
  H1N1, Day 7,30-48M[N=52,54] | 32 | 20
  H3N2, Day 7,17-29M[N=53,52] | 36 | 8
  H3N2, Day 7,30-48M[N=54,54] | 39 | 23
  Victoria, Day 7,17-29M[N=53,52] | 40 | 8
  Victoria, Day 7,30-48M[N=52,54] | 39 | 16
  Yamagata, Day 7, 17-29M[N=53,52] | 46 | 10
  Yamagata, Day 7, 30-48M[N=52,54] | 44 | 19

30. Secondary Outcome: MGI for Anti-neuraminidase Antibodies Titers Against Each of the Four Vaccine Strains After 1 Dose of Fluarix Quadrivalent Vaccine by Age Strata.
Description: MGI was defined as the fold increase in GMTs post-vaccination compared to Day 0. The vaccine strains included A/Christchurch/16/2010 (H1N1), A/Victoria/361/2011 (H3N2), B/Brisbane/60/2008 (Victoria) and B/Hubei-Wujiagang/158/2009 (Yamagata) antigens. The humoral response in terms of anti-neuraminidase antibodies for all vaccine strains were calculated by age stratum which included 17-29 months and 30-48 months age groups for both the Fluarix primed and unprimed groups.
Time Frame: At Day 7 post dose 1
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 54 | 54
Fold Increase
  H1N1, Day 7,17-29M[53,52] | 11.4 [8.2 to 15.8] | 1.5 [1.2 to 1.9]
  H1N1, Day 7,30-48M[N=52,54] | 6.0 [4.1 to 8.8] | 2.1 [1.7 to 2.7]
  H3N2, Day 7,17-29M[N=53,52] | 4.6 [3.6 to 5.8] | 1.7 [1.4 to 2.0]
  H3N2, Day 7,30-48M[N=54,54] | 5.3 [4.2 to 6.8] | 2.3 [1.9 to 2.8]
  Victoria, Day 7,17-29M[N=53,52] | 5.2 [4.3 to 6.3] | 1.5 [1.1 to 2.1]
  Victoria, Day 7,30-48M[N=52,54] | 5.1 [4.1 to 6.5] | 2.3 [1.6 to 3.4]
  Yamagata, Day 7, 17-29M[N=53,52] | 8.8 [7.2 to 10.8] | 2.2 [1.5 to 3.2]
  Yamagata, Day 7, 30-48M[N=52,54] | 8.7 [6.9 to 11.0] | 3.2 [2.3 to 4.5]

31. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Solicited local AEs assessed were pain, redness and swelling. Any = any solicited local AE reported irrespective of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness and swelling was defined as redness/swelling above 50 millimeter (mm).
Time Frame: During a 7-day (Day 0 to 6) follow-up period after first vaccination
Population: Analysis was performed on the Total Vaccinated cohort included all subjects with at least one vaccine administration documented and symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 239 | 228
Subjects
  Any Pain | 96 | 61
  Grade 3 Pain | 2 | 1
  Any Redness | 82 | 48
  Grade 3 Redness | 2 | 0
  Any Swelling | 49 | 25
  Grade 3 Swelling | 2 | 0

32. Secondary Outcome: Duration of Solicted Symptoms
Description: Duration was defined as number of days with any grade of solicted local and/or general symptoms
Time Frame: During the 7-day (Days 0-6) post-vaccination Dose 1 period
Population: Analysis was performed on the Total Vaccinated cohort included all subjects with at least one vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 96 | 61
Days
  Drowsiness | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 4.0]
  Irritability/fussiness | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of appetite | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0]
  Pain | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 5.0]
  Redness | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Swelling | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 5.0]
  Temperature | 1.0 [1.0 to 5.0] | 2.0 [1.0 to 6.0]

33. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were drowsiness, Irritability/Fussiness, loss of appetite and Temperature. Any Temperature = axillary temperature ≥37.5 degrees Celsius (°C). Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 Irritability/Fussiness = Crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = did not eat at all. Grade 3 temperature = axillary temperature > 39.0°C.
Time Frame: During the 7 days (Days 0 - 6) post dose 1 vaccination
Population: as for outcome 31
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 238 | 224
Subjects
  Any Drowsiness | 54 | 44
  Grade 3 Drowsiness | 5 | 1
  Related Drowsiness | 36 | 28
  Any Irritability/Fussiness | 77 | 59
  Grade 3 Irritability/Fussiness | 5 | 5
  Related Irritability/Fussiness | 51 | 43
  Any Loss of appetite | 51 | 46
  Grade 3 Loss of appetite | 8 | 5
  Related Loss of appetite | 31 | 31
  Any Temperature | 13 | 26
  Grade 3 Temperature | 2 | 1
  Related Temperature | 6 | 15

34. Secondary Outcome: Number of Subjects Reporting AEs With Medically Attended Visits (MAV)
Description: MAVs were defined as an AEs with a medically-attended visits i.e. prompting emergency room (ER) visits, hospitalizations or physician visits and that were not routine visits for physical examination or vaccination. Any MAV was defined as at least one MAV experienced. Grade 3 was a MAV that prevented normal activities and related was defined as a MAV assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 - Day 179)
Population: Analysis was performed on the Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 241 | 229
Subjects
  Any MAV | 149 | 130
  Grade 3 MAV | 5 | 8
  Related MAV | 0 | 1

35. Secondary Outcome: Number of Subjects Reporting Potential Immune-Mediated Diseases (pIMDs)
Description: pIMDs were defined as a subset of AEs that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have had an autoimmune aetiology. Any pIMDs= Any AEs that occured regardless of the relation with vaccination. Related pIMDs= Any pIMD assessed by the investigator as casually related to the study vaccination.
Time Frame: During the entire study period (Days 0 - 179)
Population: as for outcome 34
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 241 | 229
Subjects
  Any pIMD | 0 | 0
  Related pIMD | 0 | 0

36. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs.
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: Within 28 days (Days 0-27) after first vaccination
Population: as for outcome 34
Measure: Number; unit: Subjects
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 241 | 229
Subjects
  Any Unsolicted AEs | 66 | 66
  Grade 3 Unsolicted AEs | 6 | 7
  Related Unsolicted AEs | 5 | 3

37. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 - Day 179)
Population: as for outcome 34
Measure: Number; unit: Subjects
Groups:
- Fluarix Quadrivalent Unprimed Group: SuSubjects in this group were unprimed in the primary study 115345 (NCT01439360) and received 2 doses of Fluarix Quadrivalent vaccine at Days 0 and 28 in the current study. The vaccine was administered intramuscularly in the deltoid region of arm.
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Number analyzed (Participants) | 241 | 229
Subjects
  Any SAE(s) | 7 | 8
  Related SAE(s) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 179; Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period; Unsolicited symptoms: During the 28-day (Day 0-27) post-vaccination period.
Description: For the frequent adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Fluarix Quadrivalent Primed Group | Fluarix Quadrivalent Unprimed Group
Serious Adverse Events (participants affected / at risk) | 7/241 | 8/229
Other Adverse Events (participants affected / at risk) | 145/241 | 138/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Quadrivalent Primed Group (N=241) | Fluarix Quadrivalent Unprimed Group (N=229)
Gastroenteritis (Infections and infestations) | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lymphadenitis bacterial (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fluarix Quadrivalent Primed Group (N=241) | Fluarix Quadrivalent Unprimed Group (N=229)
Pain (General disorders) | 96/239 | 61/228
Redness (General disorders) | 82/239 | 48/228
Swelling (General disorders) | 49/239 | 25/228
Drowsiness (General disorders) | 54/238 | 44/224
Irritability/Fussiness (General disorders) | 77/238 | 59/224
Loss of Appetite (General disorders) | 51/238 | 46/224
Temperature (General disorders) | 13/238 | 26/224
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.